CLINICAL TRIAL: NCT05331885
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Efficacy and Safety of Suvratoxumab in Mechanically Ventilated Adults and Adolescents for the Prevention of Nosocomial Pneumonia
Brief Title: A Human Monoclonal Antibody Against Staphylococcus Aureus Alpha Toxin in Mechanically Ventilated Adult Subjects - 2
Acronym: SAATELLITE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to administrative reasons
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-320-003; SAATELLITE-2 (Other: COMBACTE-NET)
Record Dates: First submitted 2022-04-01; First posted 2022-04-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-01

CONDITIONS: Ventilator Associated Pneumonia; Staphylococcus Aureus
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Staphylococcal Infections | interventions — suvratoxumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, randomized, placebo-controlled, single-dose study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind, randomized, controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR-320 (Suvratoxumab) (Experimental): Participants will receive a single intravenous (IV) dose of suvratoxumab on Day 0 of the study.
  Interventions: Biological: Suvratoxumab
- Placebo (Placebo Comparator): Participants will receive a single IV dose of placebo to survatoxumab on Day 0 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Suvratoxumab — Monoclonal antibody
  Other Names: AR-320; MEDI4893
  Arms: AR-320 (Suvratoxumab)
Drug: Placebo — Placebo contains only excipients
  Arms: Placebo

SUMMARY:
Clinical trial looking at safety and efficacy of suvratoxumab in prevention of pneumonia caused by Staphylococcus aureus in high-risk patients

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled study evaluating the efficacy of a single IV dose of suvratoxumab in mechanically ventilated subjects in the ICU who are at high risk for S. aureus infections and who are currently free of active S. aureus-related disease but are colonized with S. aureus in the LRT.

ELIGIBILITY:
Inclusion Criteria:

1. Colonized with Staphylococcus aureus;
2. Expected to require prolonged intubation and mechanical ventilation, without any evidence of active pneumonia.

Exclusion Criteria:

1. Staphylococcal disease at randomisation;
2. Lung injury score consistent with pneumonia;
3. Chronic tracheostomy patients;
4. The study subject is moribund
5. Receipt of anti- S. aureus systemic antibiotics
6. Active pulmonary disease

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of nosocomial all-cause pneumonia through 30 days post dose | 30 days
  All-cause pneumonia is based on clinical, radiographic, and microbiologic criteria. The percent reduction of the incidence of (% of patients with) nosocomial all-cause pneumonia, regardless of identified etiology, following administration of study drug through 30 days post dose

SECONDARY OUTCOMES:
Number of participants with TEAE at 30 days | 30 days
  Treatment emergent adverse events (TEAE) are those adverse events (AEs, any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship) that occur or worsen during the treatment period, i.e., after the administration of study drug, through 30 days post dose
Number of participants with TESAE at 90 days | 90 days
  Treatment emergent serious adverse events (TESAE) are serious adverse events (SAEs, AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience; persistent or significant disability/incapacity; congenital anomaly) that, as TEAEs, are present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, through 90 days
Number of participants with TEAESI at 90 days | 90 days
  A TEAE of special interest (TEAESI) is an AE of scientific and medical interest specific to understanding of the study drug and may have required close monitoring and rapid communication by the investigator to the sponsor. An AESI may have been serious or non-serious. The time-frame is 90 days.
Number of Participants with Nosocomial all-cause pneumonia or death through 30 days post dose | 30 days
  All-cause pneumonia is based on clinical, radiographic, and microbiologic criteria. The percent reduction of the incidence of (% of patients with) nosocomial all-cause pneumonia, regardless of cause, or death following administration of study drug through 30 days post dose
Number of Participants with Nosocomial S. aureus pneumonia through 30 days post dose | 30 days
  S. aureus pneumonia is based on clinical, radiographic, and microbiologic criteria. The percent reduction of the incidence of (% of patients with) nosocomial S. aureus pneumonia following administration of study drug through 30 days post dose
Number of Participants with Nosocomial S. aureus pneumonia through 90 days post dose | 90 days
  S. aureus pneumonia is based on clinical, radiographic, and microbiologic criteria. The percent reduction of the incidence of (% of patients with) nosocomial S. aureus pneumonia following administration of study drug through 90 days post dose
Suvratoxumab Maximum Observed Serum Concentration (Cmax) | 90 days
  Maximum Observed Serum Concentration (Cmax) of suvratoxumab at Day 0 (Pre-dose, end of the infusion, 8 and 24 hours post dose), and on Days 7, 30 and 90. At Day 90 only for a subset of patients.
Suvratoxumab Area under the Plasma Concentration-Time Curve (AUC) | 90 days
  the area under the plasma concentration-time curve (AUC) will be measured from time 0 to Day 30 (AUC0-30), in all study subjects, and AUC from time 0 to Day 90 (AUC0-90) for a subset of subjects
Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to Suvratoxumab | 90 days
  The incidence of (number of patients with) positive anti-drug antibodies (ADA) titer to suvratoxumab will be assessed and summarized by number and percentage of subjects that are ADA positive at predose, Day 30 in all subjects and Day 90 in a subset of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Francois, MD, Principal Investigator — Centre Hospitalier Universitaire (CHU) de Limoges
Locations (27):
- Belgium (3):
  - Research Site Bel03, Haine-Saint-Paul
  - Research Site Bel02, Ottignies
  - Research Site Bel05, Yvoir
- France (9):
  - Research Site Fra05, Argenteuil
  - Research Site Fra16, La Roche-sur-Yon
  - Research Site Fra10, Le Mans
  - Research Site Fra08, Lille
  - Fra06, Limoges
  - Research Site Fra07, Orléans
  - Research Site Fra15, Pierre-Bénite
  - Research Site Fra12, Tours
  - Research Site Fra03, Trévenans
- Research Site GRC01, Larissa, Greece
- Israel (4):
  - Research Site ISR03, Haifa
  - Research Site ISR05, Holon
  - Research Site ISR01, Ramat Gan
  - Research Site ISR06, Safed
- Netherlands (3):
  - Research Site NLD01, Enschede
  - Research Site NLD03, Heerlen
  - Research Site NLD02, Utrecht
- Spain (7):
  - Research Site SPA04, Barcelona
  - Research Site SPA01, Córdoba
  - Research Site SPA07, Madrid
  - Research Site SPA08, Santander
  - Research Site SPA06, Santiago de Compostela
  - Research Site SPA03, Terrassa
  - Research Site SPA05, Valencia

IPD SHARING:
Plan to Share IPD: No